CLINICAL TRIAL: NCT06877936
Title: Determination of Scapulothoracic and Glenohumeral Angles by Imaging in Patients After Shoulder Arthroplasty
Brief Title: Determination of Scapulothoracic and Glenohumeral Angles by Imaging in Patients After Shoulder Arthroplasty (SCAP-imag)
Acronym: SCAP-imag
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ramsay Générale de Santé (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2024-A01684-43
Record Dates: First submitted 2025-03-10; First posted 2025-03-14 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Arthropathy Shoulder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Reverse total shoulder arthroplasty surgery (Experimental): Reverse total shoulder arthroplasty surgery performed by Dr. Lionel Neyton about 2 years prior to inclusion in the study
  Interventions: Procedure: EOS exam; Other: Questionnaires Constant et ASES

INTERVENTIONS:
Procedure: EOS exam — The EOS procedure will consist of taking 3 x-rays per side (6 in total) while the patient is standing (oriented at 35° to the x-ray) with the arm in position 0°, then at 45° and finally at 90° elevation in the frontal plane for 20 seconds per position.
Other: Questionnaires Constant et ASES — There will be 2 questionnaires : Constant and American Shoulder and Elbow Surgeons to determine their pain level and functional limitations.

SUMMARY:
The shoulder is a site particularly affected by osteoarthritis since it affects up to 7% of the population aged over 65. To deal with osteoarthritis, total shoulder prosthesis is an increasingly used solution. Among the different types of total shoulder prostheses, the majority of surgical procedures involve the use of a reverse total shoulder prosthesis. This type of prosthesis modifies the anatomy of the shoulder in order to ensure better stability and mobility of the shoulder in patients while also compensating for potential significant lesions of certain deep muscles of the shoulder joint (i.e., rotator cuff).

Reverse prostheses have good short-term results but these are impaired in longer term with a Constant functional score of around 70% at 10 years and a survival rate of 70% after 20 years. Problems of bone conflicts between the scapula and the humerus can also be observed on these reverse total shoulder prostheses with variable rates from 4.6% to 47.3% depending on the position of the prosthesis.

In order to minimize the risk of complications, several tools are available to surgeons to optimize the positioning of the prosthesis. Planning software can be used to plan the kinematics of the shoulder after arthroplasty and quantify shoulder movements by 1/ estimating the scapulothoracic and glenohumeral angles, and 2/ determining the scapulohumeral rhythm (i.e., joint coordination index evaluating the relative contribution of these two joints to the total elevation of the arm). This prediction allows the surgeon to adapt the size, shape and position of the implants to each patient in order to ensure optimal shoulder kinematics, namely a maximum amplitude without bone conflicts (contacts) between the scapula and the humerus.

The main objective of this study is to evaluate the influence of a reverse shoulder arthroplasty on shoulder kinematics at 2 years postoperatively in comparison with the non-operated contralateral limb.

ELIGIBILITY:
Inclusion Criteria:

* Major
* Reverse total shoulder arthroplasty surgery performed by Dr. Lionel Neyton (Jean Mermoz Private Hospital,69008 Lyon) 24±3 months prior to inclusion in the study.
* Have had a CT scan of the operated shoulder prior to the operation
* Patient having signed informed consent
* Patient affiliated to a social security scheme or beneficiary of such a scheme, according to Article L.1124-1 of the Public Health Code

Exclusion Criteria:

* Contraindication to the EOS® examination
* Anthropometry incompatible with the production of EOS images
* Pregnant, parturient, breastfeeding women
* Have a history of fracture at the level of the humerus, scapula or clavicle
* Have a history of surgery on the shoulder or contralateral upper limb to the limb with the prosthesis
* Protected patient: adult under guardianship, curatorship or other legal protection, deprived of liberty by judicial or administrative decision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-01-29 (Actual); Primary Completion 2026-01-29 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Kinematics evaluation | one month
  The evaluation of kinematics will be done through the quantification of the scapulothoracic and glenohumeral angles.

SECONDARY OUTCOMES:
Scapulohumeral rhythm | one month
  Scapulohumeral rhythm on the operated side and on the contralateral side.
Constant score on the operated side and the contralateral side. | one month
  Constant score
ASES score | one month
  ASES score on the operated side and the contralateral side.

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital privé Jean Mermoz, Lyon, France